CLINICAL TRIAL: NCT04537520
Title: Interventional Multi-Center Post Market Randomized Controlled Open-Label Clinical Trial Comparing Kerecis Omega3 Wound Versus SOC in Hard to Heal Diabetic Foot Wounds
Brief Title: Interventional Clinical Trial Comparing Kerecis Omega3 Wound Versus SOC in Diabetic Foot Wounds
Acronym: KereFish
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre d'Etudes et de Recherche pour l'Intensification du Traitement du Diabète (Other)
Collaborators: Kerecis Ltd. (Industry); RCTs (Industry); Clininfo S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-A01743-52
Record Dates: First submitted 2020-08-25; First posted 2020-09-03 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Diabetes; Diabetic Foot Ulcer
Keywords: Complex diabetic foot wounds; Kerecis Omega3Wound; extracellular matrix
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): treatment with the device Kerecis Omega3 Wound
  Interventions: Device: Kerecis Omega3 Wound
- Control Group (No Intervention): treatment with SOC treatment

INTERVENTIONS:
Device: Kerecis Omega3 Wound — Treatment of the wound with Kerecis Omega3 Wounds matrices
  Arms: Experimental Group

SUMMARY:
The KereFish study is a randomized controlled study to study the efficacy of Kerecis Omega3 Wound on deep diabetic ulcers. This study is probably the first in his field: in this one, the Kerecis Omega3 Wound dies are used on the types of wounds for which they are ultimately intended. This study aims to document the cost benefits of earlier closure of severe diabetic wounds, or the change of the deep and chronic wound into a smaller and shallower ulcer, and to radically alter its prognosis. The study, carried out in France, uses the pre-existing home nursing system with the transmission of photographs to the reference centre. The study was largely designed to ensure transparency of the financial calculations involved.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients, regardless of the age of their diabetes, with a grade UT 2 or 3 lower limb sore; grade 2: wound penetrating to the tendon or capsule. UT grade 3: wound penetrating to the bone or joint OR hospitalized/ambulatory patients for diabetic foot sores or amputations, which have not closed or are dehiscent.
* Patients who can tolerate aggressive surgical debridement
* Patients without severe ischemia IPS - 0.6 or pressure of the big toe - 50mmHg
* Longness of the wound: 30 days (does not apply to amputation wounds; patients may be included when the wound is less than 30 days old) OR if the amputation level is under the ankle
* Patients willing and able to give informed consent to participate in the clinical trial.
* Male or female over the age of 18
* Patients living at a geographical distance compatible with referral nurse visits
* Negative pregnancy test for women of childbearing age who do not use contraception.
* Patients covered by social security
* Patients who are capable (in the investigator's opinion) and willing to comply with all clinical trial requirements

Exclusion Criteria:

* Patients whose wound surface is not measurable
* Patients with unsealed osteomyelitis
* Patients with fever related to a foot infection (it may be reassessed at a later time when the infection is gone)
* Patients with a necrotic wound that will not tolerate aggressive surgical debridement
* Immunosuppressed patients
* Patients with systemic corticosteroids or other treatments that may delay wound healing
* Pregnant, breast-feeding or planning pregnancy during the clinical trial
* Any other significant disease or disorder that the investigator believes may pose a risk to participants because of their participation in the clinical trial or that may influence the outcome of the clinical trial or the participant's ability to participate in the clinical trial.
* Patients with rheumatoid arthritis
* Patients with systemic lupus
* Patients with a known skin allergy to fish
* Patients deprived of liberty by judicial or administrative decision, persons subject to a legal protection measure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2020-07-02 (Actual); Primary Completion 2022-07-09 (Actual); Study Completion 2022-12-16 (Actual)

PRIMARY OUTCOMES:
Wound area | Week 0
  measuring the surface of the wound with planimetry software
Wound area | Week 16
  measuring the surface of the wound with planimetry software

CONTACTS AND LOCATIONS:
Overall Officials: Dured DARDARI, MD, Principal Investigator — Centre Hospitalier Sud Francilien
Locations (12):
- France (12):
  - CHU de Caen, Caen
  - Centre Hospitalier Sud Francilien, Corbeil-Essonnes
  - CHU de Dijon - Bocage Sud, Dijon
  - Hotel Dieu Le Creusot, Le Creusot
  - CHU de Montpellier, Montpellier
  - Hôpital Cochin, Paris
  - Hopital Bichat-Claude Bernard, Paris
  - CHU de Reims - Hôpital Debré, Reims
  - Hôpital de Roubaix - CETRADIM, Roubaix
  - CHU de Nantes Hôpital Nord Laennec, Saint-Herblain
  - CHRU de Strasbourg - Hopital Civil, Strasbourg
  - CHU de Toulouse Hôpital Rangueil, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dardari D, Potier L, Sultan A, Francois M, M'Bemba J, Bouillet B, Chaillous L, Kessler L, Carlier A, Jalek A, Sbaa A, Orlando L, Bobony E, Detournay B, Kjartansson H, Bjorg Arsaelsdottir R, Baldursson BT, Charpentier G. Intact Fish Skin Graft vs. Standard of Care in Patients with Neuroischaemic Diabetic Foot Ulcers (KereFish Study): An International, Multicentre, Double-Blind, Randomised, Controlled Trial Study Design and Rationale. Medicina (Kaunas). 2022 Dec 1;58(12):1775. doi: 10.3390/medicina58121775. PMID 36556977